CLINICAL TRIAL: NCT02137317
Title: Prevention of Farmers' Exposure to Pesticides With Relevant Personal Protective Equipment in Chitwan District of Nepal
Brief Title: Farming, Personal Protective Equipment, Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other); Odense University Hospital (Other); Dialogos (Unknown); Nepal Development Society (Unknown); Nepal Public Health Foundation (Unknown); Nepal Red Cross Society (Unknown); Dansk Selskab for Arbejds- og Miljømedicin (Unknown); The Augustinus Foundation, Denmark. (Other); Else og Mogens Wedell Wedellsborgs Foundation (Unknown); Syngenta (Unknown); BASF (Industry)
Responsible Party: Principal Investigator, Anshu Varma, MPH, Cand.scient.san.publ, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: FAPPEN
Record Dates: First submitted 2014-05-07; First posted 2014-05-13 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Organophosphate Poisoning
Keywords: Pesticides; Personal protective equipment; Developing countries; Tropical Climate
MeSH Terms: conditions — Organophosphate Poisoning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LAPPE/DP (Experimental): In the LAPPE experiment the farmer will work as usual (mixing/loading/application/cleaning). wearing the LAPPE solution and carrying a new hand pressured backpack sprayer with a standardized nozzle. Conditions such as dosage, work practices and weather conditions will remain uncontrolled but be observed. After one week this process will be repeated wearing the DP solution.
  Interventions: Device: LAPPE (locally adapted personal protective equipment)
- DP/LAPPE (Active Comparator): In the DP experiment the farmer will work as usual (mixing/loading/application/cleaning) wearing the DP solution and carrying his usual backpack sprayer with his usual nozzle. Conditions such as dosage, work practices and weather conditions will remain uncontrolled but be observed. After one week this process will be repeated wearing the LAPPE solution.
  Interventions: Device: LAPPE (locally adapted personal protective equipment)

INTERVENTIONS:
Device: LAPPE (locally adapted personal protective equipment) — * Hand: Nitrile gloves flexible enough to grip pesticide container firmly and in a length appropriate for mixing and spraying such as wrist length. They should not contain lining inside. In case, nothing is available disposable plastic bags can provide sufficient protection. In both cases wearing a cotton glove underneath.
  * Upper and lower body: As thick or as heavy cotton blouse and trousers as can be worn and plastic sheets cut as a long poncho.
  * Feet: Unlined rubber boots or shoes at least calf height with thick cotton socks underneath with possibility for trousers to be worn outside rubber boots or shoes.

SUMMARY:
According to the World Health Organization pesticide poisoning is a major health problem due to the millions of cases annually occurring worldwide. Farmers have a particularly high risk of pesticide poisoning because of their work involving pesticide use to protect crops. The majority of pesticide poisonings occur in developing countries. On a short term it is not realistic to reduce farmers' use of pesticides significantly because it would require that secure and cost-effective alternatives are introduced. This is a lengthy process, which should undoubtedly be supported. However, it becomes as important to make sure that farmers can protect themselves from pesticide exposure meanwhile. Use of personal protective equipment can minimize pesticide exposure on farmers' bodies and consequently reduce their risk of pesticide poisoning. However, the sparse research identified through a systematic literature review shows that we are not in a position to give recommendations on what personal protective equipment farmers should protect themselves with against pesticide exposure suitable to their specific conditions. The purpose of the present study is to examine factors that influence farmers' use of personal protective equipment during their work with organophosphates and, based on this examine the ability of locally adapted personal protective equipment to reduce their organophosphate exposure. The hypothesis is that farmers working in locally adapted personal protective equipment have less acute organophosphate poisoning symptoms, a higher plasma cholinesterase level and find it to be a more feasible solution than farmers working in their daily practice wearing. Examining how locally adapted personal protective equipment (onwards referred to as the LAPPE solution) performs in practice implies testing it in an intervention study. A randomized crossover experiment design is chosen partly because fewer farmers have to be recruited since each farmer will act as his own control and partly because the between farmer variation is strongly reduced. The performance of the LAPPE solution will be tested in one experiment and compared to the performance of the same farmers' daily practice wearing (onwards referred to as the DP solution) in another experiment. The LAPPE solution is expected to have a superior performance. The participation sequence (LAPPE/DP or DP/LAPPE) will be randomized. The study will be conducted among farmers in Chitwan, Nepal.

DETAILED DESCRIPTION:
LITERATURE SEARCH STRATEGY:

Based on recommendations from information specialists in the field of health, agriculture and technology the following databases were chosen to search for scientific literature about the present study's purpose: Pubmed, Embase, SveMed, CAB abstracts (Centre for Agriculture and Biosciences International), Agris, DADS (Denmark's Technical University's Digital Library), Scopus and Ebsco. The key search terms for the literature search were: personal protective equipment, farmers, pesticides, developing countries and tropical climate. Synonyms for each of these search terms were identified by means of Gyldendals Dictionary and previous international literature. In Pubmed, SveMed, Embase, CAB abstracts and Agris the synonyms were applied to find subject headings which the main search was based on. However, in DADS, Scopus, Ebsco searches on subject headings was not an option and therefore the main search was based on the synonyms.

* Pubmed: 3349 hits, subject headings for key terms personal protective equipment and pesticides with no limitations.
* Embase: 399 hits, subject headings for key terms personal protective equipment and pesticides with the limitation human.
* SveMed: 24 hits, subject headings for key terms personal protective equipment and pesticides.
* CAB abstracts: 607 hits, subject headings for key terms personal protective equipment and pesticides.
* Agris: 681 hits, subject headings for key terms personal protective equipment and pesticides.
* DADS 8650 hits, subject headings for key terms personal protective equipment and pesticides.
* Scopus: 1988 hits, synonyms for key terms personal protective equipment and pesticides and developing countries and tropical climate with the limitation to human.
* EBSCO: 722 hits, synonyms for key terms personal protective equipment and pesticides.

Firstly, the relevance of titles was evaluated, secondly the relevance of abstracts from hits with relevant titles was evaluated and thirdly the relevance of full texts from hits with relevant abstracts was evaluated. A search was made based on the function 'related studies' for each relevant study in each database. The reference list of each relevant study was viewed and searched in Web of Science for citations. Finally each accessible relevant study was read carefully (5 hits). Exclusion criteria were studies on closed farming, mechanized farming, non-tropical conditions, and farming in industrialized countries or laboratory performance testing of personal protective equipment seeing that these criteria would not represent typical farming conditions in developing countries. Grey literature was searched in databases of the International Labor Organization, World Health Organization and Food and Agricultural Organization.

STUDY AREA:

Nepal is divided into 75 administrative districts. Pesticide consumption data show that excessive use of pesticides is common in different crops such as rice, maize, wheat and vegetables production areas. Chitwan District is selected purposively for three reasons:

* One of the highest vegetable growing districts of Nepal is Chitwan.
* An excessive pesticide use is documented in Chitwan.
* An unpublished study being the first of its kind in Nepal known to the research group documents the seriousness of the problem in Chitwan. A comparative cross-sectional study was conducted among 90 vegetable farmers using hand pressured backpack sprayers and 90 blood donors. Fifty %, 15 % and 13 % of the pesticides used by the vegetable farmers could be categorized as moderately, highly and slightly hazardous, respectively, according to the World Health Organization Hazard Classification. Organophosphates were one of the most common pesticides used by the vegetable farmers; the moderately hazardous chlorpyrifos and imidacloprid as well as the highly hazardous dichlorvos. Poor working practices without adequate safety precautions were common among the vegetable farmers. The vegetable farmers reported a higher number of acute organophosphate poisoning symptoms and had lower levels of acetyl cholinesterase than blood donors. Chitwan has a total population of around 566,661 and was a largely uncultivated dense forest before the Nepali government started spraying with the insecticide dichlorodiphenyltrichloroethane for a Malaria Eradication Project in the 1950s. Immediately, Chitwan became a major farming region and services and infrastructure expanded across the area. Out of a total 46,894 hectare of arable land, 44,291 hectare is used for agricultural purpose (maize, rice, wheat, beans, lentils, mustard and vegetables). Agriculture is the primary source of income for 75 % of the population. Around 4000-5000 people of the working population is engaged in vegetable farming. Chitwan has 40 village district committees and the District Agricultural Office considers 10 of these as pocket areas in terms of vegetable farming based on their own observations, experiments, monitoring and personal communication with vegetable farmers. The ten pocket areas are Mangalpur, Jagatpur, Shukranagar, Chainpur, Bhandara, Gitanagar, Sibanagar, Jutpani, Kumroj and Padampur. To the extent that it is possible farmers fulfilling the inclusion and exclusion criteria of the present study in these pocket areas will be recruited:

RECRUITMENT STRATEGY:

Non-probability.

SAMPLE SIZE DETERMINATION:

The sample size calculations are based on a quasi-experimental unpublished study of 25 vegetable farmers from Chitwan whose acute organophosphate poisoning symptoms and plasma cholinesterase levels were measured pre and post an organophosphate spraying session on the same day during daily practice conditions.

* Mean number of acute organophosphate poisoning symptoms 1.08±1.32 (Pre spraying measurement) 2.4±1.87 (Post spraying measurement) 0.0003 (P-value)
* Mean U/ml level of plasma cholinesterase 1.41±0.59 (Pre spraying measurement) 1.29±0.54 (Post spraying measurement) 0.0548 (P-value)

The pre and post organophosphate spraying measurements are considered to represent the "healthiest" and "unhealthiest" condition that the vegetable farmers can be expected to be in, respectively. Thus, for the present study the pre and post organophosphate spraying measurements are expected to resemble the results among the farmers after having worked with organophosphates wearing the LAPPE solution and DP solution, respectively. A sample size suitable to the study resources was gained when applying the pre and post results of the number of acute organophosphate poisoning symptoms.

* Paired means = 1.08, 2.4
* Paired standard deviations = 1.320,1.870
* Correlation = 0
* Sides = 1, 2
* Alpha = 0.05
* Power = 0.9

Taking into consideration dropouts, technical problems leading to invalid measurements, refusals and co-variables for multivariate analyses 33 % of the sample size (34 pairs) is added, the result being rounded up to 50 pairs of farmers needed for the present study.

DATA ANALYSES:

Descriptive:

* Frequency, proportion categorical variables
* Mean, minimum, maximum and standard deviation of numeric variables
* Table crossing background, explanatory and feasibility variables with LAPPE/DP experiment
* Table crossing number of acute organophosphate poisoning symptoms with plasma cholinesterase levels U/ml

Unadjusted (paired t-test and McNemar test):

* Mean difference in number of acute organophosphate poisoning symptoms after both experiments
* Mean difference in plasma cholinesterase level U/ml after both experiments

Adjusted (mixed model):

* Number of acute organophosphate poisoning symptoms after the LAPPE experiment is compared to the number of acute organophosphate poisoning symptoms after the DP experiment adjusted for baseline values, period effect, experiment sequence and explanatory variables.
* Plasma cholinesterase level U/ml after the LAPPE experiment is compared to the plasma cholinesterase level U/ml after the DP experiment adjusted for baseline values, period effect, experiment sequence and explanatory variables.

Sensitivity:

To allow confidence in the main finding its robustness will be assessed by repeating the analyses with more rigid health outcome definitions if possible such as:

* Farmers with acute organophosphate poisoning symptoms before the LAPPE and DP experiment are excluded.
* Farmers with more abnormal plasma cholinesterase levels U/ml before the LAPPE and DP experiment are excluded.
* Farmers with chronic illness are excluded.
* Farmers who respond to the "fake" symptoms are excluded.

ETHICAL CONSIDERATIONS:

Informal recognition and encouragement in Chitwan will be obtained from the District Agricultural Office and District Public Health Office. An advisory opinion from the Danish Ethics Committee will be obtained. Informed consents will be retrieved from farmers participating in the pre-testing and experiments.

The plasma cholinesterase measurement will make it possible to identify farmers with abnormal levels. If such cases occur the farmer will be excluded from the study and given advice on how to proceed. The small amount of blood required is not considered as damaging to the farmers' health. However, the finger stick may have minor risks such as momentary pain when the lancet goes into the finger, bruise, visible and sore puncture site for a short period, feeling of dizziness or light headedness. Disposable finger stick lancets will be used to avoid any infectious transmission.

The LAPPE solution will be provided to the farmers after their participation with an information folder and oral explanation on how to store the LAPPE. Despite the results of the study, the LAPPE solution is an improvement in farmers' current practice which is that they basically do not protect themselves according to the recommendations of World Health Organization or Food and Agricultural Organization.

The choice of organophosphates for the experiments will be based on the type of organophosphates that the farmers already use. In other words, the farmers will not be exposed to less or more dangerous pesticides than what they usually expose themselves to. During the data collection the organophosphates will be stored according to their safety label recommendations. In case, the remaining organophosphates cannot be used in other studies they will be disposed by taking safety precautions as recommended by the World Health Organization.

During all study activities a first aid kit will be accessible and the data collectors will wear basic personal protective equipment during the experiments and informed about a safe handling of organophosphates.

During data entry, data is stored on two external hard disks and the principal investigator's computer in the control of the principal investigator. Data on the Test Mate ChE Cholinesterase System is automatically deleted when the power is switched off. Every week a full backup of the data file will be saved on a USB stick placed outside research establishments under the principal investigator's control until the data entry is complete. Data editing and analysis will be based on a data file without sensitive information (like name, address and phone number). The data file will be saved on an external hard disk, USB stick and the principal investigator's computer drop box on a daily basis and kept under secure conditions and with only access to the principal investigator.

The following data will be stored in a locked safe under research establishments in the sole control of the principal investigator:

* Original data
* File with raw data
* File with analyzable and anonymized data
* File linking farmers' sensitive information with their study identification number

The following data will be stored in a locked safe outside research establishments in the sole control of the principal investigator and safe owners:

• File with analyzable data excluding sensitive information

If necessary, during analysis and interpretation of results the research group can get access to the file with analyzable and anonymized data through e-mail. However, the e-mail will not contain the file linking sensitive information with study identification numbers and is therefore considered as being manually encrypted.

Upon completion of the research study the original data will be cut into pieces, placed in a sealable bag which can be tightly tied, fill the bag with water and then transfer the bag to a waste container. Blood tests and materials used in this regard will be given to Nepal Red Cross Society. Data stored outside research establishments will be retrieved. Two independent data files; one file with analyzable data excluding sensitive information and another file with farmers' sensitive information linking to their study identification number and scanned copies of informed consents will be stored in Nepal for up to five years. Potential permission to store data in Denmark will be seeked from the Danish Data Protection Agency. Upon approval data will be sent to the Danish Data Archive for indefinite storage time with data documentation. The condition for data access to the Danish Data Archive is that only the principal investigator will have access to the data and full control of giving permission for sharing data with others in the future. If sharing of data occurs the new researcher will have to seek approval from the Danish Data Protection Agency and then consult the Danish Data Archive.

ELIGIBILITY:
Inclusion

* Male (females usually wear national dresses considered to provide adequate protection (43).
* Age min. 18 years (implies being a legal worker).
* Grows crops in knee and abdomen height in given data collection period.
* Willing to spend 1.5-3 hours working with organophosphates under normal working conditions.
* Involved in farming minimum two years (implies being active).
* Usually sprays at least once in two weeks with organophosphates on average (implies being active).
* Uses a hand pressured backpack sprayer placed at home (necessary to complete non-intervention).
* Works with crops in 5-10 katha land (sufficient to apply organophosphates for given time).
* Has a mobile/landline number (necessary for easy contact).

Exclusion

* Has a helper during work with organophosphates (organophosphate exposure reduced).
* Is unwilling to stay organophosphate free one week prior to each of two experiment days (necessary for comparable measurements).
* Has any of the following conditions: liver disease/damage, alcoholic/viral hepatitis, acute infection, chronic malnutrition, heart attack, metastasis, obstructive jaundice, inflammation, uses pyridostigmine drugs (decreases or increases plasma cholinesterase) (44-46).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Plasma Cholinesterase | Farmers will be followed over 15 days (cholinesterase measured four times)
  Plasma cholinesterase is a substance necessary for the proper functioning of the human nervous system. The inhibition of this type of cholinesterase is considered as a useful indicator of exposure to organophosphates when measured before and after likely exposure. Plasma cholinesterase will be measured with a Test-mate Cholinesterase System (Model 400) requiring 10 microliters (µL) for a blood test.

SECONDARY OUTCOMES:
Acute Organophosphate Poisoning Symptoms | Farmers will be followed for 15 days (symptoms measured four times)
  The World Health Organization has constructed a clinical representation of acute organophosphate poisoning consisting of: headache, dizziness, bradycardia, weakness, anxiety, excessive sweating, fasciculations, abdominal cramps, dyspnea, miosis, paralysis, salivation, tearing, ataxia, pulmonary edema, vomiting, diarrhea, confusion, acetyl cholinesterase inhibition. In the present study, all clinical representations except from acetyl cholinesterase inhibition will be evaluated as self-reported acute organophosphate poisoning symptoms. However, some of the clinical representations may be difficult for the farmers' to report themselves and therefore such clinical representations have been translated into more understandable terms. Furthermore, symptoms are added based on local health care experience. In a survey information on self-reported acute organophosphate poisoning symptoms will be retrieved with yes/no response options as has been seen in previous studies.

OTHER OUTCOMES:
Feasibility | Farmers will be followed over 15 days (measured two times)
  In the survey the feasibility of the LAPPE solution (locally adapted personal protective equipment) is measured with yes/no response options: "Was it comfortable?", "Did it feel hotter?", "Any problem when spraying?" and "Did you like garments?". With minor adjustments the same questions will be posed to the farmers in the present study to measure the feasibility of the LAPPE and DP solutions.

CONTACTS AND LOCATIONS:
Overall Officials: Anshu Varma, Principal Investigator — Bispebjerg Hospital
Locations (1):
- FAPPEN - Field, Bharatpur, Chitwan, Nepal

REFERENCES:
- [Background] 1. FAO. International Code of Conduct on the Distribution and Use of Pesticides. Rome: Food and Agriculture Organization of the United Nation, 2002.
- [Background] Thundiyil JG, Stober J, Besbelli N, Pronczuk J. Acute pesticide poisoning: a proposed classification tool. Bull World Health Organ. 2008 Mar;86(3):205-9. doi: 10.2471/blt.08.041814. PMID 18368207
- [Background] Jeyaratnam J. Acute pesticide poisoning: a major global health problem. World Health Stat Q. 1990;43(3):139-44. PMID 2238694
- [Background] Konradsen F. Acute pesticide poisoning--a global public health problem. Dan Med Bull. 2007 Feb;54(1):58-9. PMID 17349229
- [Background] 5. Fait A, Iversen B, Tiramani M, Visentin S, Maroni M. Preventing health risks from the use of pesticides in agriculture. Geneva: World Health Organization. 2001.
- [Background] 6. Acutely toxic pesticides: initial input on extent of problem and guidance for risk management. Fourth session of the Intergovernmental Forum on Chemical Safety. Doc number: IFCS/FORUM-IV/10w; April 2003.
- [Background] 7. Epidemiology of pesticide poisoning: harmonized collection of data on human pesticide exposure in selected countries. Geneva: International Programme on Chemical Safety/WHO; 2004.
- [Background] Konradsen F, van der Hoek W, Cole DC, Hutchinson G, Daisley H, Singh S, Eddleston M. Reducing acute poisoning in developing countries--options for restricting the availability of pesticides. Toxicology. 2003 Nov 5;192(2-3):249-61. doi: 10.1016/s0300-483x(03)00339-1. PMID 14580791
- [Background] Atreya K, Sitaula BK, Overgaard H, Bajracharya RM, Sharma S. Knowledge, attitude and practices of pesticide use and acetylcholinesterase depression among farm workers in Nepal. Int J Environ Health Res. 2012;22(5):401-15. doi: 10.1080/09603123.2011.650154. Epub 2012 Jan 24. PMID 22273496
- [Background] Bhanti M, Shukla G, Taneja A. Contamination levels of organochlorine pesticides and farmers' knowledge, perception, practices in rural India: a case study. Bull Environ Contam Toxicol. 2004 Nov;73(5):787-93. doi: 10.1007/s00128-004-0496-8. No abstract available. PMID 15669720
- [Background] Gomes J, Lloyd O, Revitt DM, Norman JN. Erythrocyte cholinesterase activity levels in desert farm workers. Occup Med (Lond). 1997 Feb;47(2):90-4. doi: 10.1093/occmed/47.2.90. PMID 9156478
- [Background] Gomes J, Lloyd OL, Revitt DM. The influence of personal protection, environmental hygiene and exposure to pesticides on the health of immigrant farm workers in a desert country. Int Arch Occup Environ Health. 1999 Jan;72(1):40-5. doi: 10.1007/s004200050332. PMID 10029229
- [Background] Jors E, Morant RC, Aguilar GC, Huici O, Lander F, Baelum J, Konradsen F. Occupational pesticide intoxications among farmers in Bolivia: a cross-sectional study. Environ Health. 2006 Apr 21;5:10. doi: 10.1186/1476-069X-5-10. PMID 16630337
- [Background] Karunamoorthi K, Mohammed A, Jemal Z. Peasant association member's knowledge, attitudes, and practices towards safe use of pesticide management. Am J Ind Med. 2011 Dec;54(12):965-70. doi: 10.1002/ajim.21008. Epub 2011 Sep 14. PMID 21919031
- [Background] Khan DA, Shabbir S, Majid M, Ahad K, Naqvi TA, Khan FA. Risk assessment of pesticide exposure on health of Pakistani tobacco farmers. J Expo Sci Environ Epidemiol. 2010 Mar;20(2):196-204. doi: 10.1038/jes.2009.13. Epub 2009 Jun 17. PMID 19536076
- [Background] 16. Matthews GA. Attitudes and behaviours regarding use of crop protection products-A survey of more than 8500 smallholders in 26 countries. Crop Prot. 2008: 27:834-846.
- [Background] Ntow WJ, Gijzen HJ, Kelderman P, Drechsel P. Farmer perceptions and pesticide use practices in vegetable production in Ghana. Pest Manag Sci. 2006 Apr;62(4):356-65. doi: 10.1002/ps.1178. PMID 16532443
- [Background] Palis FG, Flor RJ, Warburton H, Hossain M. Our farmers at risk: behaviour and belief system in pesticide safety. J Public Health (Oxf). 2006 Mar;28(1):43-8. doi: 10.1093/pubmed/fdi066. Epub 2006 Jan 25. PMID 16436451
- [Background] Oliveira Pasiani J, Torres P, Roniery Silva J, Diniz BZ, Dutra Caldas E. Knowledge, attitudes, practices and biomonitoring of farmers and residents exposed to pesticides in Brazil. Int J Environ Res Public Health. 2012 Aug 24;9(9):3051-68. doi: 10.3390/ijerph9093051. PMID 23202670
- [Background] Plianbangchang P, Jetiyanon K, Wittaya-Areekul S. Pesticide use patterns among small-scale farmers: a case study from Phitsanulok, Thailand. Southeast Asian J Trop Med Public Health. 2009 Mar;40(2):401-10. PMID 19323025
- [Background] Recena MC, Caldas ED, Pires DX, Pontes ER. Pesticides exposure in Culturama, Brazil--knowledge, attitudes, and practices. Environ Res. 2006 Oct;102(2):230-6. doi: 10.1016/j.envres.2006.01.007. Epub 2006 Feb 21. PMID 16497291
- [Background] Salameh PR, Baldi I, Brochard P, Abi Saleh B. Pesticides in Lebanon: a knowledge, attitude, and practice study. Environ Res. 2004 Jan;94(1):1-6. doi: 10.1016/s0013-9351(03)00092-6. PMID 14643280
- [Background] 23. Shrestha P, Koirala P, Tamrakar AS. Knowledge, practice and use of pesticides among commerical vegetable growers of Dhading district, Nepal. The Journal of Agriculture and Environment. 2010;11:95--100.
- [Background] Singh B, Gupta MK. Pattern of use of personal protective equipments and measures during application of pesticides by agricultural workers in a rural area of Ahmednagar district, India. Indian J Occup Environ Med. 2009 Dec;13(3):127-30. doi: 10.4103/0019-5278.58915. PMID 20442830
- [Background] Sivayoganathan C, Gnanachandran S, Lewis J, Fernando M. Protective measure use and symptoms among agropesticide applicators in Sri Lanka. Soc Sci Med. 1995 Feb;40(4):431-6. doi: 10.1016/0277-9536(94)00143-h. PMID 7725116
- [Background] Sosan MB, Akingbohungbe AE. Occupational insecticide exposure and perception of safety measures among cacao farmers in southwestern Nigeria. Arch Environ Occup Health. 2009 Fall;64(3):185-93. doi: 10.1080/19338240903241077. PMID 19864221
- [Background] Yassin MM, Abu Mourad TA, Safi JM. Knowledge, attitude, practice, and toxicity symptoms associated with pesticide use among farm workers in the Gaza Strip. Occup Environ Med. 2002 Jun;59(6):387-93. doi: 10.1136/oem.59.6.387. PMID 12040114
- [Background] Chester G, Adam AV, Inkmann Koch A, Litchfield MH, Tuinman CP. Field evaluation of protective equipment for pesticide operators in a tropical climate. Med Lav. 1990 Nov-Dec;81(6):480-8. PMID 2100762
- [Background] 29. Lee SA, Yang SC. Studies on contamination patterns, penetration of pesticides through clothing and spray operator protection. The Planter 1991;67(778):9-40.
- [Background] Machado-Neto JG, Matuo T, Matuo YK. Semiquantitative evaluation of dermal exposure to granulated insecticides in coffee (Coffea arabica L.) crop and efficiency of individual protective equipment. Bull Environ Contam Toxicol. 1996 Dec;57(6):946-51. doi: 10.1007/s001289900281. No abstract available. PMID 8875843
- [Background] 31. Shaw A, Nomula R, Patel B. Protective clothing and application control for pesticide applicators in India: A field study. ASTM special technical publication 2000;342-53.
- [Background] 32. Shaw A. Field evaluation of protective clothing worn by pesticide applicators in hot climates. International Pest Control 2008;May/June:152-5.
- [Background] Keifer MC. Effectiveness of interventions in reducing pesticide overexposure and poisonings. Am J Prev Med. 2000 May;18(4 Suppl):80-9. doi: 10.1016/s0749-3797(00)00144-6. PMID 10793284
- [Background] 34. Neupane D. Pesticides exposure and its health effects among commercial vegetable farmers in Nepal. (unpublished dissertation). Esbjerg: University of Southern Denmark; 2012.
- [Background] 35. Pesticide Registration and Management Section. Annual Report. Plant Protection Directorate, Department of Agriculture, Haribhawan. Lalitpur: Nepal.2009;pp.41.
- [Background] 36. Agri-business Promotion and Statistics Division. Statistical information on Nepalese agriculture 2007/08. Government of Nepal, 2008.
- [Background] 37. World Health Organization. The WHO recommended classifications of pesticides by hazard and guidelines to classification 2009. World Health Organization. Geneva: Switzerland. 2010.
- [Background] Yabiku ST, Schlabach S. Social Change and the Relationships between Education and Employment. Popul Res Policy Rev. 2009 Aug 1;28(4):533-549. doi: 10.1007/s11113-008-9117-2. PMID 21461188
- [Background] 39. Axinn WG, Yabiku ST. Social change, the social organization or families, and fertility limitation. American Journal of Sociology. 2001;106:1219-61.
- [Background] 40. Shivakoti GP, Axinn WG, Bhandari P, Chehetri N. The impact of community context on land use in an agricultural society. Population and Environment. 1999;20(3):191-213.
- [Background] 41. District Agricultural Office. Chitwan: District Agriculture Office; 2011.
- [Background] 42. National Library of Medicine. Pubmed Health. A.D.A.M. Medical Encyclopedia. Last reviewed: May 28, 2013. Cholinesterase.
- [Background] 43. EQM Research I. Test-mate cholinesterase test system Instruction Manual. 2003. Available from: www.eqmresearch.com.
- [Background] 44. EQM Research I. Description of the test-mate CHE. 2012. Available from: www.eqmresearch.com.
- [Background] Catano HC, Carranza E, Huamani C, Hernandez AF. Plasma cholinesterase levels and health symptoms in peruvian farm workers exposed to organophosphate pesticides. Arch Environ Contam Toxicol. 2008 Jul;55(1):153-9. doi: 10.1007/s00244-007-9095-0. Epub 2007 Dec 19. PMID 18157496
- [Background] 46. Encyclopedia of Occupational Health and Safety. 2012. Cholinesterase. www.ilo.org/oshenc.
- [Background] Kapka-Skrzypczak L, Cyranka M, Skrzypczak M, Kruszewski M. Biomonitoring and biomarkers of organophosphate pesticides exposure - state of the art. Ann Agric Environ Med. 2011;18(2):294-303. PMID 22216802
- [Background] Hofmann JN, Carden A, Fenske RA, Ruark HE, Keifer MC. Evaluation of a clinic-based cholinesterase test kit for the Washington State Cholinesterase Monitoring Program. Am J Ind Med. 2008 Jul;51(7):532-8. doi: 10.1002/ajim.20588. PMID 18459125
- [Background] Rajapakse BN, Thiermann H, Eyer P, Worek F, Bowe SJ, Dawson AH, Buckley NA. Evaluation of the Test-mate ChE (cholinesterase) field kit in acute organophosphorus poisoning. Ann Emerg Med. 2011 Dec;58(6):559-564.e6. doi: 10.1016/j.annemergmed.2011.07.014. PMID 22098995
- [Background] 50. Food and Agricultural Organization. Guidelines for personal protection when working with pesticides in tropical climates. Rome: Food and Agricultural Organization; 1990.
- [Derived] Varma A, Neupane D, Ellekilde Bonde JP, Jors E. Is prevention of acute pesticide poisoning effective and efficient, with Locally Adapted Personal Protective Equipment? A randomized crossover study among farmers in Chitwan, Nepal. Med Lav. 2016 Jul 26;107(4):271-83. PMID 27464900